CLINICAL TRIAL: NCT04727450
Title: Effects of Multimodal Training of Combined Cognitive and Physical and Cognitive or Physical Training Only on Cognition and Physical Fitness of Older Adults: A Cluster Randomized Controlled Trial
Brief Title: Effects of Multimodal Training of Combined Cognitive and/or Physical Training on Cognition and Fitness of Older Adults
Acronym: MTCCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Jacobs University Bremen gGmbH (Other); The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Chow Bik-chu, Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 12607620
Record Dates: First submitted 2021-01-17; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Cognitive Decline; Cognitive Impairment, Mild
Keywords: Intervention programs; Older adults; Cognitive & Physical Training; Cluster RCT; Multimodal
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training; Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: Cluster RCT. Each elderly center as a cluster will be randomly assigned to be either an intervention group (IG) to receive intervention training modes (A: cognitive training, B: physical training only, C: CCPT) or a control group (CG). IGs will either receive integrated format of ABC or two training modes of AB or BC or CA.
Who Masked: Outcomes Assessor
Masking Description: No information will be given to test administrators about intervention or control groups with the exception of project staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1. Integrated format (Active Comparator): Integrated or Combination of ABC of A: cognitive training. B: physical training and C: Combined Cognitive and Physical Training (CCPT).
  Interventions: Behavioral: Cognitive training; Behavioral: physical training; Behavioral: Combination of cognitive and physical training (CCPT)-BIGMAP
- 2. Cognitive training + Physical Training (A+B) (Active Comparator): Intervention of A & B treatments.
  Interventions: Behavioral: Cognitive training; Behavioral: physical training
- 3. Physical training + CCPT (B+C) (Active Comparator): Intervention of B & C treatments.
  Interventions: Behavioral: physical training; Behavioral: Combination of cognitive and physical training (CCPT)-BIGMAP
- 4. CCPT + Cognitive training (C+A) (Active Comparator): Intervention of C & A treatments.
  Interventions: Behavioral: Cognitive training; Behavioral: Combination of cognitive and physical training (CCPT)-BIGMAP
- 5. Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Cognitive training — Involves participants engaging in selected games which require thinking skills to be played in a group of 2-4 people.
  Arms: 1. Integrated format; 2. Cognitive training + Physical Training (A+B); 4. CCPT + Cognitive training (C+A)
Behavioral: physical training — Involves learning of preselected routines of "line dancing" taught by a line dance instructor.
  Arms: 1. Integrated format; 2. Cognitive training + Physical Training (A+B); 3. Physical training + CCPT (B+C)
Behavioral: Combination of cognitive and physical training (CCPT)-BIGMAP — BIGMAP is a program engaging participants in specially designed cognitive/memory games together with physical training (Fu & Chow, 2019).
  Other Names: "Brain Invigoration Gross Motor Activation Program" (BIGMAP)
  Arms: 1. Integrated format; 3. Physical training + CCPT (B+C); 4. CCPT + Cognitive training (C+A)

SUMMARY:
The elderly population worldwide is expected to increase exponentially. There will be a higher percentage of older adults suffering cognitive decline in the coming decades. Cognitive impairment, being the most common health problem associated with ageing, contributes to possible loss of functional independence and disability. The purpose of this study is to determine the effectiveness of four mixed modalities of three training programs (combined cognitive and physical training [CCPT], cognitive or physical training only) on cognition and fitness of community-dwelling older adults in Hong Kong. The study hypotheses will be set as the integrated format of all three training will have higher cognition and fitness scores than other combinations of two training modes and all these mixed modalities will have greater positive outcomes than the active control subjects.

DETAILED DESCRIPTION:
The study design is a cluster randomized controlled trial. Twenty-four elderly centers as clusters will be randomly selected and assigned to be intervention (n=20) or control groups (n=4) in two study phases. A total of 8-10 older adults (age ≥ 60) from each cluster (total subjects = 228) will be invited to be study participants. Each intervention cluster will receive either an integrated training format or one out of three combinations of two training modes. Each intervention training mode will last for 2-month of 16 sessions in total, 2 sessions per week and 60 min per session, hence, the total intervention will last for 4 months for two training modes or an integrated training format. Assessments will be conducted at pre-test, two post-training tests, and a 2-month follow-up test after completion of all training.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 or above
2. Both gender
3. Willingness and capability to participate in this study and training
4. Willingness and capability to give informed consent to participate in this study
5. Pass the cutting-point of referenced screening tests (cognitive and emotional)

Screening tools:

* MOCA score above 19 (satisfactory basic function)
* Positive and Negative Syndrome Scale (PANSS) with scores < 19 in positive scale, < 22 in negative scale, and < 38 in general psychopathology scale

Exclusion Criteria:

1. A history of systematic cardiovascular diseases, poorly controlled hypertension, stroke, Parkinson's disease
2. Early stages of Alzheimer's Disease, or the use of psychoactive drugs
3. Complicated conditions that preclude regular attendance of the training
4. Currently receiving regular physical (perform aerobic, flexibility and stretching exercises for 3 days per week, 45 minutes per session, for 1 year or longer) and cognitive exercises (such as playing mahjong, chess, bridge and reading for more than 30 minutes per session and 3 times per week, for 1 year or longer ).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Tests: for executive function (pre-test) | Pre-test (1st test): before intervention
  Wisconsin Card Sorting Test (WCST) for the executive function will be conducted (20-30 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.
Cognitive Tests: for executive function (2nd test) | 2nd test: after 2-month intervention
  Wisconsin Card Sorting Test (WCST) for the executive function will be conducted (20-30 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.
Cognitive Tests: for executive function (3rd test) | 3rd test: after 4-month intervention
  Wisconsin Card Sorting Test (WCST) for the executive function will be conducted (20-30 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.
Cognitive Tests: for executive function (4th test) | 4th test: after 2-month follow up
  Wisconsin Card Sorting Test (WCST) for the executive function will be conducted (20-30 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.
Cognitive Tests: for attention (pre-test) | Pre-test (1st test): before intervention
  Color Trail Making test (CTMT) for attention will be conducted (5-8 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.
Cognitive Tests: for attention (2nd test) | 2nd test: after 2-month intervention
  Color Trail Making test (CTMT) for attention will be conducted (5-8 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.
Cognitive Tests: for attention (3rd test) | 3rd test: after 4-month intervention
  Color Trail Making test (CTMT) for attention will be conducted (5-8 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.
Cognitive Tests: for attention (4th test) | 4th test: after 2-month follow up
  Color Trail Making test (CTMT) for attention will be conducted (5-8 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.
Cognitive Tests: for everyday memory (pre-test) | Pre-test (1st test): before intervention
  Rivermead Behavioral Memory Test (RBMT) for everyday memory will be conducted (30 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.
Cognitive Tests: for everyday memory (2nd test) | 2nd test: after 2-month intervention
  Rivermead Behavioral Memory Test (RBMT) for everyday memory will be conducted (30 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.
Cognitive Tests: for everyday memory (3rd test) | 3rd test: after 4-month intervention
  Rivermead Behavioral Memory Test (RBMT) for everyday memory will be conducted (30 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.
Cognitive Tests: for everyday memory (4th test) | 4th test: after 2-month follow up
  Rivermead Behavioral Memory Test (RBMT) for everyday memory will be conducted (30 min, unit on a scale) in four evaluation time frames, respectively. The evaluators at all sessions will be blind to the group membership of participants.

SECONDARY OUTCOMES:
Fitness Tests: BMI (pre-test) | Pre-test (1st test): before intervention
  Weight and height will be tested and combined to report BMI in kg/m^2 in four evaluation time frames
Fitness Tests: BMI (2nd test) | 2nd test: after 2-month intervention
  Weight and height will be tested and combined to report BMI in kg/m^2 in four evaluation time frames
Fitness Tests: BMI (3rd test) | 3rd test: after 4-month intervention
  Weight and height will be tested and combined to report BMI in kg/m^2 in four evaluation time frames
Fitness Tests: BMI (4th test) | 4th test: after 2-month follow up
  Weight and height will be tested and combined to report BMI in kg/m^2 in four evaluation time frames
Fitness Tests: Senior physical fitness test battery (pre-test) | Pre-test (1st test): before intervention
  Senior physical fitness test
Fitness Tests: Senior physical fitness test battery (2nd test) | 2nd test: after 2-month intervention
  Senior physical fitness test
Fitness Tests: Senior physical fitness test battery (3rd test) | 3rd test: after 4-month intervention
  Senior physical fitness test
Fitness Tests: Senior physical fitness test battery (4th test) | 4th test: after 2-month follow up
  Senior physical fitness test
Four square step test for dynamic balance (pre-test) | Pre-test (1st test): before intervention
  Four square step test
Four square step test for dynamic balance (2nd test) | 2nd test: after 2-month intervention
  Four square step test
Four square step test for dynamic balance (3rd test) | 3rd test: after 4-month intervention
  Four square step test
Four square step test for dynamic balance (4th test) | 4th test: after 2-month follow up
  Four square step test

OTHER OUTCOMES:
Behavioral and motivation survey (pre-test) | Pre-test (1st test): before intervention
  Survey on motivation and subjective health status rating
Behavioral and motivation survey (2nd test) | 2nd test: after 2-month intervention
  Survey on motivation and subjective health status rating
Behavioral and motivation survey (3rd test) | 3rd test: after 4-month intervention
  Survey on motivation and subjective health status rating
Behavioral and Motivation Survey (4th test) | 4th test: after 2-month follow up
  Survey on motivation and subjective health status rating
Depression and Loneliness Survey (pre-test) | Pre-test (1st test): before intervention
  The Center for Epidemiological Studies-Depression scale (CES-D) and Loneliness
Depression and Loneliness Survey (2nd test) | 2nd test: after 2-month intervention
  The Center for Epidemiological Studies-Depression scale (CES-D) and Loneliness
Depression and Loneliness Survey (3rd test) | 3rd test: after 4-month intervention
  The Center for Epidemiological Studies-Depression scale (CES-D) and Loneliness
Depression and Loneliness Survey (4th test) | 4th test: after 2-month follow up
  The Center for Epidemiological Studies-Depression scale (CES-D) and Loneliness
Physical activity participation Survey (pre-test) | Pre-test (1st test): before intervention
  Physical activity participation (TTM)
Physical activity participation Survey (2nd test) | 2nd test: after 2-month intervention
  Physical activity participation (TTM)
Physical activity participation Survey (3rd test) | 3rd test: after 4-month intervention
  Physical activity participation (TTM)
Physical activity participation Survey (4th test) | 4th test: after 2-month follow up
  Physical activity participation (TTM)

CONTACTS AND LOCATIONS:
Overall Officials: Bik-Chu CHOW, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Hong Kong Baptist University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
In our application of university human ethics, we have declared non-disclosure of individual data.

REFERENCES:
- [Background] Fu F, Chow BC. Brain Invigoration and Gross Motor Activation Programme (BIGMAP). Hong Kong Baptist University, Hong Kong. 2019. ISBN: 9789881542137
- [Derived] Chow BC, Jiao J, Man D, Lippke S. Study protocol for 'the effects of multimodal training of cognitive and/or physical functions on cognition and physical fitness of older adults: a cluster randomized controlled trial'. BMC Geriatr. 2022 May 6;22(1):398. doi: 10.1186/s12877-022-03031-5. PMID 35524188